CLINICAL TRIAL: NCT06911606
Title: A Prospective Phase II Clinical Study of Serplulimab Combined With Platinum-containing Doublet Induction Therapy for Limited-stage Small Cell Lung Cancer (LS-SCLC) Followed by Surgery or Radiotherapy
Brief Title: Study of Serplulimab Plus Chemotherapy as Neoadjuvant Therapy for Limited-stage Small Cell Lung Cancer (LS-SCLC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: Liaoning Cancer Hospital & Institute (Other); Guangzhou No.12 People's Hospital (Other Government); Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Wen-zhao ZHONG, Principal Investigator, Clinical Professor, Guangdong Provincial People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLX10IIT110; HLX10IIT110 (Other: Guangdong Provincial People's Hospital)
Record Dates: First submitted 2025-03-10; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: SCLC, Limited Stage
Keywords: II-IIIB (N2) LS-SCLC
MeSH Terms: interventions — Etoposide; Carboplatin; Cisplatin; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 4 cycles of Serplulima plus platinum-containing dual drug (Experimental): After 4 cycles of Serplulimab combined with etoposide and carboplatin or cisplatin then MDT determines surgery or radical radiotherapy
  Interventions: Drug: 4 cycles of Serplulimab combined with etoposide and carboplatin or cisplatin

INTERVENTIONS:
Drug: 4 cycles of Serplulimab combined with etoposide and carboplatin or cisplatin — After 4 cycles of Serplulimab combined with etoposide and carboplatin or cisplatin then MDT determines surgery or radical radiotherapy
  Other Names: surgery

SUMMARY:
This investigator-initiated, open-label, prospective Phase II clinical trial, planned to take place across multiple centers in China. We aimed to evaluate the efficacy and safety of surgical resection or chemotherapy following serplulimab plus platinum-containing dual induction therapy for stage II-IIIB (N2) LS-SCLC

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in clinical research and sign written informed consent
2. Male or female patients aged 18-75 years old (including the critical value)
3. Histologically or cytologically confirmed SCLC
4. Clinically diagnosed as IIB-IIIB ( N2) stage (AJCC 8th edition cancer staging)
5. Patients who have not received systemic anti-tumor treatment or chest radiotherapy in the past
6. By Surgeons evaluate patients who have no contraindications to surgery
7. According to Response Evaluation Criteria in Solid Tumors (RECIST 1.1), there is at least one radiologically measurable lesion
8. ECOG score 0-1
9. Expected survival time > 6 months
10. Hepatitis B surface antigen (HBsAg) (-) and hepatitis B core antibody (HBcAb) (-). If HBsAg (+) or HBcAb (+), the hepatitis B virus deoxyribonucleic acid (HBV-DNA) must be <2500 copies/mL or 500 IU/mL before inclusion. Subjects who are HCV antibody (-) or HCV-RNA negative can be enrolled if HCV-RNA is positive, the subject must have alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤ Only 3×ULN can join the group. Subjects who are co-infected with hepatitis B and hepatitis C need to be excluded (positive HBsAg or HBcAb test, and positive HCV antibody test)
11. Laboratory tests within 7 days before the first use of the study drug confirm sufficient organ and bone marrow function, No serious hematopoietic abnormalities, cardiac, liver, renal dysfunction or immune deficiency (no blood transfusion, albumin, recombinant human thrombopoietin or colony-stimulating factor (CSF) treatment within 14 days before the first medication in this study)
12. Female patients must meet one of the following conditions: a. Menopause (defined as the absence of menstruation for at least 1 year without other confirmed reasons other than menopause), or b. Have undergone surgical sterilization (removal of ovaries and/or uterus) , or c. Have childbearing potential, but must meet the following requirements: the serum/urine pregnancy test within 7 days before enrollment must be negative, and agree to use contraceptive measures with an annual failure rate of <1% or maintain abstinence (avoiding heterosexual intercourse) (from signing ICF to at least 6 months after the last dose of study drug) (contraceptive methods with annual failure rates <1% include bilateral fallopian tube ligation, male sterilization, correct use of hormonal contraceptives that inhibit ovulation, and hormone-releasing intrauterine contraception devices and copper-containing IUDs or condoms), and you must not breastfeed.
13. Male patients must meet the following requirements: Agree to abstain from sex (avoid heterosexual intercourse) or take contraceptive measures, as follows: When the partner is a female of childbearing age or the partner is pregnant, the male patient must agree to abstain from sexual intercourse (avoiding heterosexual intercourse) or take contraceptive measures for at least 6 months during the study treatment period and after the last dose of the study drug. Maintain abstinence or use condoms during the first trimester to prevent embryonic drug exposure. Periodic abstinence (for example, calendar days, ovulation period, basal body temperature or post-ovulation contraceptive method) and in vitro ejaculation are unqualified contraceptive methods
14. The end of previous non-systemic anti-tumor treatment must be ≥ 2 weeks from the start of medication, and according to Common Terminology Criteria for Adverse Events (CTCAE) 5.0, treatment-related AEs reverted to grade ≤1 (except grade 2 alopecia).

Exclusion Criteria:

1. Mixed SCLC confirmed by histology or cytology
2. Previously received systemic anti-tumor treatment for small cell lung cancer, including but not limited to chemotherapy, immunotherapy, and radiotherapy
3. Other active malignant tumors within 5 years or at the same time. Cured localized tumors, such as basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, carcinoma in situ of the prostate, carcinoma in situ of the cervix, and carcinoma in situ of the breast, can be enrolled
4. Those who are planning to undergo or have received organs in the past or bone marrow transplant patients
5. Pleural effusion, pericardial effusion or ascites requiring clinical intervention
6. Myocardial infarction or poorly controlled arrhythmia (including men with QTc interval) within 6 months before the first administration of the study drug ≥450 ms, women ≥470 ms) (QTc interval is calculated by Fridericia's formula)
7. The subject has uncontrolled or symptomatic hypercalcemia (> 1.5 mmol/L ionized calcium or calcium > 12 mg/dL or Corrected serum calcium > ULN)
8. The patient has grade ≥ 2 CTCAE peripheral neuropathy
9. Human immunodeficiency virus (HIV) infection, HIV antibody test results are positive
10. Suffering from active pulmonary tuberculosis
11. Past and There are currently subjects with interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, severely impaired lung function, etc. who are judged by the researcher to be likely to interfere with the detection and treatment of suspected drug-related pulmonary toxicity
12. Hepatitis B (HBsAg or HBcAb test is positive, and HBV-DNA test is positive), Hepatitis C (HCV antibody test is positive, and HCV-RNA test is positive). Subjects with co-infection of hepatitis B and hepatitis C (positive HBsAg or HBcAb test, and positive HCV antibody test). Note: Hepatitis B patients who have been stabilized by antiviral treatment (HBV-DNA ≤ 2500 copies/mL or 500IU/mL) can be enrolled
13. Subjects have known active or suspected autoimmune diseases. Subjects who are in stable condition and do not require systemic immunosuppressant treatment are allowed to enroll
14. Those who have received live vaccine treatment within 28 days before the first dose. However, inactivated viral vaccines are allowed to treat seasonal influenza, but intranasal live attenuated influenza vaccines are not allowed
15. Systemic corticosteroids (> 10 mg/ subjects treated with prednisone effective doses) or other immunosuppressive drugs. However, the following conditions are allowed: in the absence of active autoimmune disease, subjects are allowed to use topical or inhaled steroids and adrenal hormone replacement therapy at a dose of ≤ 10 mg/day prednisone effective dose
16. Any active infection requiring systemic anti-infectious therapy within 14 days before study drug administration, or the subject has a positive RT-PCR test for SARS-CoV-2 infection at enrollment. Subjects with a history of COVID-19 infection must have a negative RT-PCR test before the first administration of the study drug
17. Have undergone major surgery within 28 days before the first administration of the study drug. The definition of major surgery in this study: at least 3 weeks of recovery time are required after surgery before the surgery can be treated in this study
18. The subject has previously received other antibodies/drugs targeting immune checkpoints, such as PD-1, PD -L1, CTLA-4 and other treatments
19. Are participating in other interventional clinical studies, or plan to start treatment in this study less than 28 days from the end of treatment in a previous interventional clinical study
20. Known to have a risk for any monoclonal antibody History of severe allergies
21. Known allergic reaction to carboplatin/cisplatin or etoposide components
22. Pregnant or lactating women
23. Subjects known to have a history of psychotropic drug abuse or drug use
24. According to the researcher's judgment, the subject has other factors that may cause the study to be terminated early.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-05-22 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
pathological complete response rate | Within 2 weeks after radical surgery
  The proportion of residual tumor cells evaluated under the microscope by the pathologist

SECONDARY OUTCOMES:
Objective response rate | Once every 2 cycles(each cycle is 21 days) during the combined treatment phase
  Measured according to RECIST1.1 evaluation criteria
Event-free survival | Follow-up at the end of cycle 2(each cycle is 28 days), 3 to 5 weeks after the last chemotherapy, 30 days after surgery, every 3 months within two years from enrollment or until death
  Assess whether the lesion is operable and measure the progression of the lesion according to the RECIST1.1 assessment criteria
Overall survival | Follow-up every 3 months and every 6 months within two years from enrollment or until death
  Lesions were measured according to RECIST1.1 evaluation criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China